CLINICAL TRIAL: NCT02196077
Title: A Randomized, Double Blind, Chronic Dosing (28 Days), Four Period, Five Treatment, Incomplete Block, Multi Center, Crossover Study to Assess the Efficacy and Safety of PT009, PT008, and PT005 in Subjects With Moderate to Severe COPD
Brief Title: Efficacy and Safety Study of PT009, PT008, and PT005 in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: PT009001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PT009001
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Budesonide and formoterol inhalation aerosol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BFF MDI 320/9.6 μg (Experimental): Budesonide and formoterol fumarate metered dose inhaler (BFF MDI) 320/9.6 μg; PT009 administered as 2 inhalations, twice daily (BID)
  Interventions: Drug: BFF MDI 320/9.6 μg
- BFF MDI 160/9.6 μg (Experimental): Budesonide and formoterol fumarate metered dose inhaler (BFF MDI)160/9.6 μg; PT009 administered as 2 inhalations, twice daily (BID)
  Interventions: Drug: BFF MDI 160/9.6 μg
- BFF MDI 80/9.6 μg (Experimental): Budesonide and formoterol fumarate metered dose inhaler (BFF MDI) 80/9.6 μg; PT009 administered as 2 inhalations, twice daily (BID)
  Interventions: Drug: BFF MDI 80/9.6 μg
- BD MDI 320 μg (Experimental): Budesonide metered dose inhaler (BD MDI) 320 μg; PT008 administered as 2 inhalations, twice daily (BID)
  Interventions: Drug: BD MDI 320 μg
- FF MDI 9.6 μg (Experimental): Formoterol fumarate metered dose inhaler (FF MDI) 9.6 μg; PT005 administered as 2 inhalations, twice daily (BID)
  Interventions: Drug: FF MDI 9.6 μg

INTERVENTIONS:
Drug: BFF MDI 320/9.6 μg — Budesonide and formoterol fumarate metered dose inhaler (BFF MDI) 320/9.6 μg; PT009 administered as 2 inhalations, twice daily (BID)
  Arms: BFF MDI 320/9.6 μg
Drug: BFF MDI 160/9.6 μg — Budesonide and formoterol fumarate metered dose inhaler (BFF MDI) 160/9.6 μg; PT009 administered as 2 inhalations, twice daily (BID)
  Arms: BFF MDI 160/9.6 μg
Drug: BFF MDI 80/9.6 μg — Budesonide and formoterol fumarate metered dose inhaler (BFF MDI) 80/9.6 μg; PT009 administered as 2 inhalations, twice daily (BID)
  Arms: BFF MDI 80/9.6 μg
Drug: BD MDI 320 μg — Budesonide metered dose inhaler (BD MDI) 320 μg; PT008 administered as 2 inhalations, twice daily (BID)
  Arms: BD MDI 320 μg
Drug: FF MDI 9.6 μg — Formoterol fumarate metered dose inhaler (FF MDI) 9.6 μg; PT005 administered as 2 inhalations, twice daily (BID)
  Arms: FF MDI 9.6 μg

SUMMARY:
This is a Phase IIb, randomized, double blind, chronic dosing (28 days), four period, five treatment, incomplete block, crossover design in subjects with moderate to severe COPD. The overall objective is to demonstrate that the combination of budesonide (BD; PT008) and formoterol fumarate (FF; PT005) in a metered-dose inhaler (MDI); (BFF MDI; PT009) provides benefit on lung function compared with BD MDI in subjects with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form (ICF) prior to any study related procedures
* COPD Diagnosis: Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Tobacco Use: Current or former smokers with a history of at least 10 pack years of cigarette smoking
* Women of non-childbearing potential or medically acceptable contraception for women of child-bearing potential and males with female partners of childbearing potential
* Severity of Disease: Subjects with an established clinical history of COPD and severity defined as: FEV1/forced vital capacity (FVC) ratio of <0.70; At Screening (Visit 1a/b), post bronchodilator FEV1 must be <80% predicted normal value, calculated using NHANES III (Third National Health and Nutrition Examination Survey) reference equations; the measured FEV1 must also be ≥30% of predicted normal value; at Visit 2, the average of the 60 minutes and 30 minutes pre dose FEV1 assessments must be <80% predicted normal value calculated using NHANES III reference equations
* Screening clinical laboratory tests must be acceptable to the Investigator
* Screening ECG must be acceptable to the Investigator
* Chest x ray or computerized tomography (CT) scan within 6 months prior to Visit 1a must be acceptable to the Investigator.

Exclusion Criteria:

* Significant diseases other than COPD, ie., disease or condition which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study
* Pregnancy, nursing female subjects, or subjects trying to conceive, or not using medically acceptable form of contraception
* Asthma: Subjects who have a primary diagnosis of asthma (Note: Subjects with a prior history of asthma are eligible if COPD is currently their primary diagnosis).
* Alpha 1 Antitrypsin Deficiency: Subjects who have alpha 1 antitrypsin deficiency as the cause of COPD -Active pulmonary disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, primary pulmonary hypertension, interstitial lung disease, and uncontrolled sleep apnea (ie., in the opinion of the Investigator severity of the disorder would impact the conduct of the study)-
* Clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematological, psychiatric, or other medical illness that would interfere with participation in this study
* Poorly Controlled COPD
* History of ECG abnormalities
* Cancer not in complete remission for at least 5 years
* Clinically significant, symptomatic prostatic hypertrophy
* Male subjects with a trans-urethral resection of the prostate or full resection of the prostate within 6 months prior to Screening
* Clinically significant bladder neck obstruction or urinary retention
* Inadequately treated glaucoma
* History of an allergic reaction or hypersensitivity to any drug or to any component of the formulations used in this study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Siddiqui, MD, MHSA, Study Director — Pearl Therapeutics, Inc.
Locations (17):
- United States (17):
  - Pearl Investigative Site, Rolling Hills Estates, California
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Panama City, Florida
  - Pearl Investigative Site, Tampa, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Edina, Minnesota
  - Pearl Investigative Site, Minneapolis, Minnesota
  - Pearl Investigative Site, Woodbury, Minnesota
  - Pearl Investigative Site, Saint Charles, Missouri
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Cincinnati, Ohio
  - Pearl Investigative Site, Columbus, Ohio
  - Pearl Investigative Site, Dublin, Ohio
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, Easley, South Carolina
  - Pearl Investigative Site, Greenville, South Carolina
  - Pearl Investigative Site, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4145&filename=PT009001-Protocol_Redacted_11APR2018.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 20 sites in the United States from August 2014 to March 2015. Study participation was a maximum of 28 days.
Pre-assignment Details: A Randomized, Double-Blind, Chronic Dosing (28 Days), Four-Period, Five-Treatment, Incomplete Block, Multi-Center, Crossover Study. Subjects completed final visit procedures. Final telephone follow-up occurred between 7 to 14 days from Visit 13. By-sequence tabulations of the data were not pre-specified.
Period: Overall Study
Arm/Group | Subjects
Started | 180
BFF MDI 320/9.6 μg | 155
BFF MDI 160/9.6 μg | 106
BFF MDI 80/9.6 μg | 103
BD MDI 320 μg | 108
FF MDI 9.6 μg | 157
Completed | 133
Not Completed | 47
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 14
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 24

BASELINE CHARACTERISTICS:
Population: The ITT population used in participant flow, Population is defined as all subjects who were randomized to treatment and received at least one dose of BFF MDI 320/9.6 ug, BFF MDI 160/9.6 ug, BFF MDI 80/9.6 ug, BD MDI 320 ug or FF MDI 9.6 ug. Statistical tabulations and analyses will be by randomized treatment.
Arm/Group | Subjects
Number analyzed (Participants) | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 84

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-12 on Day 29
Description: Change from Baseline in forced expiratory volume in 1 second (FEV1) area under the curve from 0 to 12 hours (AUC0-12)
Time Frame: Day 29
Population: MITT Population is a subset of the ITT population which includes subjects who received treatment and had post-treatment efficacy data from at least two Treatment Periods.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- BFF MDI 320/9.6 ug: BFF MDI 320/9.6 ug
- BFF MDI 160/9.6 ug: BFF MDI 160/9.6 ug
- BFF MDI 80/9.6 ug: BFF MDI 80/9.6 ug
- BD MDI 320 ug: BD MDI 320 ug
- FF MDI 9.6 ug: FF MDI 9.6 ug
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 148 | 98 | 96 | 99 | 142
Liters | 0.231 [0.197 to 0.266] | 0.197 [0.158 to 0.236] | 0.205 [0.165 to 0.244] | 0.011 [-0.028 to 0.050] | 0.176 [0.141 to 0.210]

2. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 Over 28 Days
Time Frame: Over 28 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 151 | 100 | 97 | 102 | 147
Liters | 0.138 [0.111 to 0.165] | 0.121 [0.089 to 0.153] | 0.110 [0.078 to 0.142] | 0.022 [-0.009 to 0.054] | 0.083 [0.056 to 0.110]

3. Secondary Outcome: Peak Change From Baseline in FEV1 (in Liters) Day 15
Time Frame: Day 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 151 | 100 | 97 | 101 | 146
Liters | 0.388 [0.354 to 0.422] | 0.366 [0.327 to 0.405] | 0.348 [0.308 to 0.387] | 0.143 [0.104 to 0.182] | 0.320 [0.286 to 0.354]

4. Secondary Outcome: Peak Change From Baseline in FEV1 (in Liters) Day 29
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 148 | 98 | 96 | 99 | 142
Liters | 0.390 [0.356 to 0.424] | 0.356 [0.317 to 0.395] | 0.359 [0.319 to 0.398] | 0.138 [0.099 to 0.177] | 0.322 [0.287 to 0.356]

5. Secondary Outcome: Peak Change From Baseline in FEV1 on Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 151 | 100 | 97 | 104 | 148
Liters | 0.338 [0.304 to 0.372] | 0.310 [0.271 to 0.349] | 0.314 [0.275 to 0.354] | 0.096 [0.058 to 0.135] | 0.313 [0.279 to 0.347]

6. Secondary Outcome: Forced Vital Capacity (FVC) AUC0-12 on Day 29
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 148 | 98 | 96 | 99 | 142
Liters | 0.305 [0.244 to 0.365] | 0.245 [0.176 to 0.315] | 0.267 [0.196 to 0.337] | 0.002 [-0.068 to 0.071] | 0.253 [0.191 to 0.314]

7. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score on Day 29
Description: Min/Max Range of TDI scale -9 (major deterioration) to +9 (major improvement)
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Full Range); unit: Index
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 149 | 97 | 96 | 100 | 142
Index | 0.598 [0.298 to 0.899] | 0.882 [0.518 to 1.246] | 0.459 [0.093 to 0.825] | -0.109 [-0.468 to 0.250] | 0.260 [-0.047 to 0.566]

8. Secondary Outcome: Change From Baseline in Average Daily Use of Rescue Ventolin HFA Over the Last Week of Treatment
Time Frame: Visit 12-13 (7 days)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 152 | 101 | 98 | 104 | 149
Puffs | 0.05 [-0.34 to 0.43] | 0.16 [-0.27 to 0.58] | 0.24 [-0.19 to 0.67] | 0.96 [0.54 to 1.38] | 0.44 [0.06 to 0.83]

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time subjects received their first dose of study medication, during the entire study period, and up to 14 days from the date of the last study medication dose.
Description: The Safety population was defined as all subjects who were randomized to treatment and received at least 1 dose of the study treatment. Subjects in the Safety population were analyzed according to the treatment received.
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | BFF MDI 80/9.6 ug | BD MDI 320 ug | FF MDI 9.6 ug
Serious Adverse Events (participants affected / at risk) | 4/155 | 2/106 | 3/103 | 4/108 | 2/157
Other Adverse Events (participants affected / at risk) | 12/155 | 2/106 | 5/103 | 8/108 | 8/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 320/9.6 ug (N=155) | BFF MDI 160/9.6 ug (N=106) | BFF MDI 80/9.6 ug (N=103) | BD MDI 320 ug (N=108) | FF MDI 9.6 ug (N=157)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 320/9.6 ug (N=155) | BFF MDI 160/9.6 ug (N=106) | BFF MDI 80/9.6 ug (N=103) | BD MDI 320 ug (N=108) | FF MDI 9.6 ug (N=157)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
Hypertension (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.